CLINICAL TRIAL: NCT04626258
Title: A Randomized Controlled Trial to Compare the Efficacy of a Medical Grade Honey Formulation (L-Mesitran®) and Fluconazol (Diflucan®) for the Treatment of Recurrent Vulvovaginal Candidiasis
Brief Title: Fluconazol Versus Medical Honey in the Treatment of Recurrent Vulvovaginal Candidiasis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL 73794.068.20
Record Dates: First submitted 2020-10-23; First posted 2020-11-12 (Actual); Last update posted 2020-11-12 (Actual); Status verified 2020-10

CONDITIONS: Candidiasis, Vulvovaginal; Recurrent Candidiasis of Vagina
Keywords: Treatment; L-Mesitran; Fluconazol; Vaginal swabs
MeSH Terms: conditions — Candidiasis, Vulvovaginal | interventions — Fluconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active comparator: Fluconazol (Active Comparator): Once a month one capsule Fluconazol 150 mg
  Interventions: Drug: Fluconazole
- L-Mesitran (Experimental): The first month every day apply L-mesitran, the next five months apply L-mesitran every week on the vagina
  Interventions: Other: L-Mesitran

INTERVENTIONS:
Drug: Fluconazole — Fluconazol once a month 150 mg capsule
  Other Names: Diflucan
  Arms: Active comparator: Fluconazol
Other: L-Mesitran — The first month apply every day one sachet, the next five months apply every week one sachet.
  Other Names: Medical honey
  Arms: L-Mesitran

SUMMARY:
The purpose of this study is to compare the efficacy of Flucanzol versus L-mesitran in the treatment of patients with recurrent vulvovaginal candidiasis. The investigator will look at vaginal swabs after 1, 6 and 12 months. The investigator included 252 patients.

ELIGIBILITY:
Inclusion Criteria:

* • Women of at least 18 years old

  * Recurrent vulvovaginal candidiasis (At least 3 episodes of clinical symptoms during the last year)
  * Clinical and microbiological diagnosis of (recurrent) vulvovaginal candidiasis at time of consultation
  * Capacity to understand, consent, and comply with the trial procedures

Exclusion Criteria:

* Mixed vaginal infections

  * Pregnancy or the intention to become pregnant during the study period
  * Women using systemic or topical antifungal medication during the last 2 weeks prior to inclusion
  * Known allergies for Fluconazole or honey
  * Candida with resistance for Fluconazole

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 252 (Estimated)
Dates: Start 2021-03-01 (Estimated); Primary Completion 2024-03-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Vaginal swab | 1 month
  The main study parameter is the mycological cure rate after one month of therapy for both the treatment (L-Mesitran®) and control (Diflucan®) groups.
Vaginal swab | 6 months
  The main study parameter is the mycological cure rate after one month of therapy for both the treatment (L-Mesitran®) and control (Diflucan®) groups.
Vaginal swab | 12 months
  The main study parameter is the mycological cure rate after one month of therapy for both the treatment (L-Mesitran®) and control (Diflucan®) groups.

SECONDARY OUTCOMES:
Quality of life will be termined with questionnaires | 1 month
  The secondary objectives are to investigate the effects of both treatments on the clinical cure rate and symptoms, including redness, irritation, itching, dysuria, dyspareunia, vaginal discharge after 1, 6, 9, and 12 months of therapy. In addition, the prophylactic activity after 6 months maintenance therapy, and the long-term efficacy as number of relapses within 12 months will be investigated. Moreover, information about side effects, discomfort, quality of life, therapy compliance, and cost of treatments for both products will be collected and compared. They will reach from no complaints-a little bit-moderate-severe
Quality of life will be termined with questionnaires | 6 months
  The secondary objectives are to investigate the effects of both treatments on the clinical cure rate and symptoms, including redness, irritation, itching, dysuria, dyspareunia, vaginal discharge after 1, 6, 9, and 12 months of therapy. In addition, the prophylactic activity after 6 months maintenance therapy, and the long-term efficacy as number of relapses within 12 months will be investigated. Moreover, information about side effects, discomfort, quality of life, therapy compliance, and cost of treatments for both products will be collected and compared.
Quality of life will be termined with questionnaires | 9 months
  The secondary objectives are to investigate the effects of both treatments on the clinical cure rate and symptoms, including redness, irritation, itching, dysuria, dyspareunia, vaginal discharge after 1, 6, 9, and 12 months of therapy. In addition, the prophylactic activity after 6 months maintenance therapy, and the long-term efficacy as number of relapses within 12 months will be investigated. Moreover, information about side effects, discomfort, quality of life, therapy compliance, and cost of treatments for both products will be collected and compared.
Quality of life will be termined with questionnaires | 12 months
  The secondary objectives are to investigate the effects of both treatments on the clinical cure rate and symptoms, including redness, irritation, itching, dysuria, dyspareunia, vaginal discharge after 1, 6, 9, and 12 months of therapy. In addition, the prophylactic activity after 6 months maintenance therapy, and the long-term efficacy as number of relapses within 12 months will be investigated. Moreover, information about side effects, discomfort, quality of life, therapy compliance, and cost of treatments for both products will be collected and compared.
Side effect of medication will be termined with questionnaires | 1 month
  The secondary objectives are to investigate the effects of both treatments on the clinicalcure rate and symptoms, including redness, irritation, itching, dysuria, dyspareunia, vaginal discharge after 1, 6, 9, and 12 months of therapy. In addition, the prophylactic activity after 6 months maintenance therapy, and the long-term efficacy as number of relapses within 12 months will be investigated. Moreover, information about side effects, discomfort, quality of life, therapy compliance, and cost of treatments for both products will be collected and compared.
Side effect of medication will be termined with questionnaires | 6 months
  The secondary objectives are to investigate the effects of both treatments on the clinicalcure rate and symptoms, including redness, irritation, itching, dysuria, dyspareunia, vaginal discharge after 1, 6, 9, and 12 months of therapy. In addition, the prophylactic activity after 6 months maintenance therapy, and the long-term efficacy as number of relapses within 12 months will be investigated. Moreover, information about side effects, discomfort, quality of life, therapy compliance, and cost of treatments for both products will be collected and compared.
Side effect of medication will be termined with questionnaires | 9 months
  The secondary objectives are to investigate the effects of both treatments on the clinicalcure rate and symptoms, including redness, irritation, itching, dysuria, dyspareunia, vaginal discharge after 1, 6, 9, and 12 months of therapy. In addition, the prophylactic activity after 6 months maintenance therapy, and the long-term efficacy as number of relapses within 12 months will be investigated. Moreover, information about side effects, discomfort, quality of life, therapy compliance, and cost of treatments for both products will be collected and compared.
Side effect of medication will be termined with questionnaires | 12 months
  The secondary objectives are to investigate the effects of both treatments on the clinicalcure rate and symptoms, including redness, irritation, itching, dysuria, dyspareunia, vaginal discharge after 1, 6, 9, and 12 months of therapy. In addition, the prophylactic activity after 6 months maintenance therapy, and the long-term efficacy as number of relapses within 12 months will be investigated. Moreover, information about side effects, discomfort, quality of life, therapy compliance, and cost of treatments for both products will be collected and compared.